CLINICAL TRIAL: NCT02635451
Title: The Relation Between Serum Ascorbic Acid Concentration and Preterm Premature Rupture of Membranes
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Mohamed Hussein Mostafa, Assistant Professor of Obstetric and Gynecology, Ain Shams Maternity Hospital
Other Study IDs: MHMostafa
Record Dates: First submitted 2015-12-15; First posted 2015-12-18 (Estimated); Last update posted 2015-12-18 (Estimated); Status verified 2015-12

CONDITIONS: Preterm Premature Rupture of Membranes
Keywords: vitamin c; Preterm Premature Rupture of Membranes
MeSH Terms: conditions — Preterm Premature Rupture of the Membranes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- study group: Study group included 20 pregnant women with PPROM and fulfilled the inclusion and exclusion criteria.
- control group: Control group also included 20 pregnant women without PPROM following every recorded case of PPROM and matched for gestational age.

SUMMARY:
To study the association between maternal serum vitamin C concentration in women with preterm premature rupture of membranes (PPROM) and women without PPROM.

DETAILED DESCRIPTION:
The micronutrient vitamin C is an effective water soluble antioxidant that scavenges several reactive oxygen species, thus reducing oxidative stress, It also acts as an enzymatic cofactor to the enzymes lysyl hydroxylase and prolyl hydroxylase, which is required for synthesis of hydroxyproline and hydroxylysine, Collagen requires hydroxyproline bridges across the triple helix to provide stability to it, Ascorbic acid also causes down regulation of the metalloproteinase-2 and biosynthesis of collagen where it is required for the formation of triple helical structure of collagen. Thus, ascorbic acid participates in the equilibrium between synthesis and degradation of collagen and this may be critical in reducing the occurrence of preterm PROM.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancies
* Gestational age between 28-37 weeks
* Rupture of membranes will be diagnosed by history, sterile speculum examination to confirm fluid leakage from the cervical canal

Exclusion Criteria:

* Patients with multiple pregnancies
* Smoker
* Polyhydramnios
* Maternal diseases such as: anemia, diabetes, UTI, RTI and vaginal infection
* History of PPROM in previous pregnancies
* Evidence of chorioamnionitis in current pregnancy

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This study will be conducted at the department of Obstetrics and Gynecology recruiting pregnant women selected from the attendees of antenatal clinic, emergency department and from inpatient wards of Ain Shams University Maternity Hospital starting from January 2016.
  This study will include 40 pregnant women between 28-37 weeks were recruited.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2016-01; Primary Completion 2016-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
relation between serum vitamin C concentration and PPROM | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Sherif M Habib, MD, Study Director — Professor of Obstetric and Gynecology